CLINICAL TRIAL: NCT01777867
Title: Pilot Studies Evaluating Cough Reflex Sensitivity and Bronchial Hyper-responsiveness: The Road to Cough and Wheeze in Patients With Gastroesophageal Reflux.
Brief Title: Cough Reflex Sensitivity and Bronchial Hyper-responsiveness
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Kenneth R. DeVault, M.D., Professor, College of Medicine, Mayo Clinic
Other Study IDs: 11-006873
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Gastroesophageal Reflux Disease; Chronic Cough; Broncho-hyperreactivity
MeSH Terms: conditions — Gastroesophageal Reflux; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Subjects in this arm were healthy volunteers. Subjects underwent both Cough Reflex Sensitivity and the Methacholine Challenge procedures.
  Interventions: Procedure: Cough Reflex Sensitivity; Procedure: Methacholine Challenge
- Non-erosive reflux disease with reflux: Subjects enrolled in this arm had non-erosive reflux disease with reflux (heartburn) for at least 6 of the preceding 12 months. Subjects underwent both Cough Reflex Sensitivity and the Methacholine Challenge procedures.
  Interventions: Procedure: Cough Reflex Sensitivity; Procedure: Methacholine Challenge
- Non-erosive reflux disease without reflux: Subjects enrolled in this arm had non-erosive reflux disease with normal levels of reflux (heartburn). Subjects underwent both Cough Reflex Sensitivity and the Methacholine Challenge procedures.
  Interventions: Procedure: Cough Reflex Sensitivity; Procedure: Methacholine Challenge

INTERVENTIONS:
Procedure: Cough Reflex Sensitivity — Subjects inhaled increasing concentrations of citric acid, which induces coughing in a dose-dependent, reproducible matter. Following each inhalation, the number of coughs in the subsequent 15 seconds was counted and recorded. The challenge was terminated once the citric acid induced 5 or more coughs and the logarithmic (base 10) concentration provoking 5 coughs was recorded.
Procedure: Methacholine Challenge — A baseline spirometry was used to assess how well the participant's lungs work by measuring how much air was inhale, how much was exhale and how quickly the participant exhaled. If this was normal, the subject inhaled slowly and deeply the methacholine test solution from a nebulizer and was told to hold their breath for 5 seconds. This was repeated until 5 inhalations were performed in no more than two minutes.

SUMMARY:
The aim of this study is to provide pilot data on the possible gastrointestinal predictors of respiratory hyper-responsiveness and how these relate to the clinical sub-types of gastroesophageal reflux disease (GERD) and visceral acid hypersensitivity.

DETAILED DESCRIPTION:
This study recruited participants into three groups: reflux patients with non-erosive disease (NERD) with abnormal levels of acid reflux, NERD patients with normal levels of reflux and healthy volunteers. Participants were assessed for cough reflex sensitivity (CRS) to citric acid and bronchial-hyperresponsiveness (BHR) to methacholine challenge, both before (baseline) and after esophageal acid infusion (HCl, 0.15M) or normal saline control (8ml/min). The order of CRS and BHR was randomized, as was the order of the acid/saline infusions.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic reflux (i.e., one symptom at least one day a week, with at least 'moderate' severity)
* no evidence of esophagitis
* non-smokers

Exclusion Criteria:

* previous gastrointestinal surgery (excluding minor surgeries, such as cholecystectomy, appendectomy
* active peptic ulcer disease
* Zollinger Ellison Syndrome
* Barrett's esophagus
* eosinophilic esophagitis
* cardiac disease
* diabetes or neurological deficit
* use of tricyclics
* selective serotonin reuptake inhibitors
* narcotics or benzodiazepines
* current use of medications that may affect symptoms of perception,lower esophageal sphincter basal pressure, acid clearance time or acid suppression
* antibiotics within 60 days
* Nursing mothers will be excluded
* allergies to citrus
* asthma
* chronic lung disease
* heart attack or stroke within the last three months
* hypersensitivity to methacholine products
* know aortic aneurysm
* uncontrolled hypertension (defined as systolic pressure greater than 200 or diastolic greater than 100)
* reduced pulmonary function test (forced expiratory volume in one second (FEV1) or the FEV1 to forced vital capacity (FVC) ratio (FEV1/FVC) of less that 70% of predicted value)
* None of the controls will have any GERD symptoms or ever used antireflux treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will recruit participants into three groups ages 18-60 years: 12 reflux patients with non-erosive disease (NERD) with abnormal levels of acid reflux, 12 NERD patients with normal levels of reflux and 12 healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in cough reflex sensitivity (CRS) | baseline, approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R. DeVault, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No